CLINICAL TRIAL: NCT05895058
Title: Comparison of 2D 4K vs. 3D HD Laparoscopic Imaging Systems in Bariatric Surgery: a Randomized Controlled Prospective Trial
Brief Title: 2D 4K vs. 3D HD in Bariatric Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marko Kraljevic (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Marko Kraljevic, PD Dr. med., Clarunis - Universitäres Bauchzentrum Basel
Organization: Clarunis - Universitäres Bauchzentrum Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D4K
Record Dates: First submitted 2023-05-14; First posted 2023-06-08 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopy
Keywords: Laparoscopy; 2D 4K vision system; 3D HD vision system; Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2D 4K laparoscopic imaging system (Experimental): Performing gastric bypass surgery intervention using a 2D 4K laparoscopic imaging system.
  Interventions: Device: Gastric bypass surgery with 2D 4K laparoscopic imaging
- 3D HD laparoscopic imaging system (Active Comparator): Performing gastric bypass surgery intervention using a 3D HD laparoscopic imaging system.
  Interventions: Device: Gastric bypass surgery with 3D HD laparoscopic imaging

INTERVENTIONS:
Device: Gastric bypass surgery with 2D 4K laparoscopic imaging — All patients involved in the investigation will receive a laparoscopic Roux-en-Y gastric bypass (LRYGB). The interventions are performed by three defined surgeons.
  Arms: 2D 4K laparoscopic imaging system
Device: Gastric bypass surgery with 3D HD laparoscopic imaging — All patients involved in the investigation will receive a laparoscopic Roux-en-Y gastric bypass (LRYGB). The interventions are performed by three defined surgeons.
  Arms: 3D HD laparoscopic imaging system

SUMMARY:
Laparoscopy has become an indispensable part of modern surgery. Vision is an important and defining element of laparoscopy and significantly affects the outcome of an operation in regard to time, mistakes and precision. Several new imaging systems have become available for laparoscopic surgery, including three-dimensional (3D) high-definition (HD), and two-dimensional (2D) ultra-high-resolution (4K) monitors. In experimental and clinical settings, several studies have been published in recent years suggesting that 3D systems present a number of potential benefits for surgeons and patients compared to the conventional 2D systems. The 3D HD system significantly reduces operation time and blood loss, and additionally shortens hospital stay. However, the performance of 3D systems against the new, ultra-high-definition 4K systems is barely known and highly controversial. There is a paucity of studies comparing these two imaging systems in clinical settings. The goal of this clinical trial is to compare 2D 4K versus 3D HD imaging systems in a complex bariatric surgery, more precisely a gastric bypass operation. The investigators aim to investigate the hypothesis stating that the use of the 3D HD system yields a significant improvement in operating time compared to a 2D 4K system in bariatric laparoscopic surgery. Furthermore, in order to give a comprehensive overview of the comparison of 2D 4K and 3D HD laparoscopy in a clinical setting, the investigators will assess the workload of the surgeon as well as the intraoperative and postoperative complications including the hospitalization time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the indication for gastric bypass according to SMOB guidelines: BMI > 35, Age > 18 and Cumulative two years of controlled conservative dieting without weight loss
* Informed Consent signed by the patient

Exclusion Criteria:

* Patients who do not have an indication for gastric bypass due to one or more of the criteria listed here: BMI > 50, Lack of adequate weight loss therapy for two years, Malignant disease, Liver cirrhosis Child A, Morbus Crohn, Carcinoma patients, Serious mental illness requiring treatment (not attributable to obesity), Chronic abuse of drugs, Lack of compliance (missed appointments, inability to cooperate), Lack of understanding of the requirements and conditions of postoperative therapy and treatment (confirmed by the specialist)
* Patient does not sign Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Operation time | intraoperative
  Operation time (OT) is defined from the beginning of the operation by incision of the skin to the end of the operation by the end of the skin suture.

SECONDARY OUTCOMES:
Intraoperative Complications | Immediately after surgery up to one day postoperatively
  Intraoperative complications are evaluated descriptively with the surgeon's documentation in the operation report and are also evaluated quantitatively according to blood loss in milliliters. Additionally, if indicated in case of intraoperative complications, a postoperative Hb control is obtained and the Hb decrease determined.
Workload of the operating surgeon | Immediately after surgery
  The condition of the operating surgeon has a great influence on the outcome of an operation. Especially when using 3D imaging, some undesirable side effects have been reported. In order to determine this once again with modern imaging and performance of a more complex procedure, it is important to determine the subjective workload of the operator. Directly after each operation performed, the operator fills out the Surg-TLX questionnaire, a validated multidimensional surgery-specific workload measure.
Postoperative Complications | Follow-up until the first postoperative Check-up after three months
  Postoperative complications are influenced by many factors, including operative time and intraoperative complications. It is important to capture these in order to also compare the postoperative outcomes of the two imaging systems. Postoperative complications are classified and documented until the first follow-up check (after three months postoperatively) in degrees I-V according to the widely used and internationally accepted Clavien Dindo Classification. In addition, the duration of hospitalization is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Kraljevic, PD Dr. med., Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel
Locations (1):
- Clarunis University Center for Gastrointestinal and Liver Diseases, Basel, Switzerland

REFERENCES:
- [Derived] Zwimpfer TA, Stiegeler N, Muller PC, Schotzau A, Fellmann-Fischer B, Heinzelmann-Schwarz V, Peterli R, Kraljevic M. Comparison of 2D 4K vs. 3D HD laparoscopic imaging systems in bariatric surgery: study protocol for a randomized controlled prospective trial. Trials. 2024 Feb 22;25(1):140. doi: 10.1186/s13063-024-07983-4. PMID 38389113